CLINICAL TRIAL: NCT00080535
Title: A Phase II Clinical Trial of Anti-Tac(Fv)-PE38 (LMB-2) Immunotoxin for Treatment of CD25 Positive Cutaneous T-Cell Lymphomas
Brief Title: Anti-Tac(Fv)-PE38 (LMB-2) to Treat Cutaneous T-Cell Lymphomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Robert Kreitman, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 040142; 04-C-0142; NCT00085085 (obsolete NCT alias)
Record Dates: First submitted 2004-04-07; First posted 2004-04-07 (Estimated); Results first posted 2012-10-24 (Estimated); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Lymphoma; T-Cell; Cutaneous
Keywords: LMB-2; Cutaneous T Cell Lymphoma; CTCL; Immunotoxin; Oncology
MeSH Terms: conditions — Lymphoma; Lymphoma, T-Cell, Cutaneous; Neoplasms | interventions — B3(Fv)-PE38KDEL recombinant immunotoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LMB-2 for cutaneous Tcell lymphoma (Experimental): 30 micrograms/kg every other day (QOD) x 3 every 4 weeks in patients with cutaneous T-cell lymphoma, a group of lymphoproliferative disorders characterized by malignant CD4+ T-lymphocytes which localize tot he skin on initial presentation.
  Interventions: Biological: LMB-2

INTERVENTIONS:
Biological: LMB-2 — 30 micrograms/kg every other day (QOD) x 3 every 4 weeks

SUMMARY:
This study will evaluate the effectiveness of an experimental drug called LMB-2 for treating cutaneous T-cell lymphoma in patients who have a protein called cluster of differentiation 25 (CD25) on their cancer cells. LMB-2 is a recombinant immunotoxin. It is made up of two parts: a genetically engineered monoclonal antibody that binds to CD25, and a toxin produced by bacteria that kills the cancer cells to which it binds. LMB-2 has killed CD25-containing cells in laboratory experiments and has caused tumors in mice to shrink. Preliminary studies in humans have shown some effectiveness in shrinking tumors in patients with various types of lymph and blood cancers.

Patients 18 years of age and older with stage 1b to IV cutaneous T-cell lymphoma that has progressed within 2 years of systemic or topical therapy and who have CD25 receptor proteins on their cancer cells may be eligible for this study. Candidates are screened with a medical history and physical examination, blood and urine tests, electrocardiogram (EKG), echocardiogram, chest x-ray, computed tomography (CT) scans of the chest, abdomen and pelvis, skin punch biopsy to evaluate tumor infiltration in the skin, and a bone marrow biopsy on patients with stage IIa disease and higher. In addition, the patient's blood, bone marrow, tumor, or other tissue is tested to determine the presence of CD25 on cancer cells.

Participants receive up to nine cycles of LMB-2 therapy as long as their cancer does not worsen and they do not develop serious side effects. Each 28-day cycle consists of 30-minute infusions of LMB-2 on cycle days 1, 3, and 5. The drug is infused through an intravenous (IV) catheter (plastic tube placed in a vein) or a central venous line - an IV tube placed in a large vein in the neck or chest that leads to the heart. In addition to drug therapy, patients undergo the following procedures:

Blood draws: Blood is drawn before, during, and after each LMB-2 infusion to measure blood levels of the drug, evaluate its effects on the cancer cells, and monitor side effects. Blood tests are also done before and during each cycle to determine how the immune system is interacting with the drug.

Disease evaluations: Patients undergo a careful skin examination, blood tests, chest x-ray, and EKG before each treatment cycle and at follow-up visits. A CT scan and echocardiogram (heart ultrasound) are done before the first cycle. Before the first and second cycles, patients have a biopsy of the lymphoma on the skin. If the biopsy is helpful in evaluating the disease response to LMB-2, additional biopsies may be requested prior to other cycles as well. A nuclear medicine scan may be done, and a bone marrow biopsy may be done in patients with stage II to IV disease. If these tests are helpful in understanding the response of the lymphoma to treatment, they may also be repeated prior to other cycles, with the patient's permission.

Patients are admitted to the National Institutes of Health (NIH) Clinical Center for the first treatment cycle. Subsequent cycles are given as outpatients. If the infusions are well tolerated, patients may return home after about one week (or possibly longer if complications occur). After returning home, patients have blood tests done weekly by their local physicians.

DETAILED DESCRIPTION:
Background:

It is estimated that 40-50% of patients with cutaneous T-cell lymphoma (CTCL) have tumors that express cluster of differentiation 25 (CD25) (Tac or IL2Ra). Normal resting T-cells do not express CD25. LMB-2 is an anti-CD25 recombinant immunotoxin containing variable domains of MAb anti-Tac and truncated Pseudomonas exotoxin. A phase I trial at National Cancer Institute (NCI) found that the maximum tolerated dose (MTD) of LMB-2 was 40 microg/Kg intravenous (IV) given every other day for 3 doses (QOD times 3) with prophylactic IV fluid. The most common adverse events were transient fever, hypoalbuminemia and transaminase elevations. In that trial, two of two patients with cutaneous T-cell lymphoma had clinical benefit (1 partial response (PR), 1 stable disease (SD)). In 1999 another recombinant fusion protein, denileukin diftitox, was approved by the Food and Drug Administration (FDA) for treatment of patients with advanced or recurrent CTCL expressing the high affinity interleukin-2 (IL-2) receptor. This receptor is composed of three subunits: CD25, CD122 and CD132. Because LMB-2 is cytotoxic to cells expressing CD25 without the other IL-2 receptor subunits needed to form the high affinity receptor, CD25+ CTCL patients are good candidates for further testing with LMB-2.

Objectives:

The purpose of this study is to determine the activity of anti-Tac(Fv)-PE38 (LMB-2) in patients with Tac-expressing Cutaneous T-cell Lymphoma (CTCL). The primary endpoints of this trial are the response rate and response duration. We will also evaluate LMB-2 immunogenicity, pharmacokinetics, and toxicity, and monitor soluble Tac levels in the serum. These will be evaluated using routine hematologic and clinical evaluation, and when appropriate, by monitoring the phenotype of circulating T-cells or of biopsied tissues using antibodies to CD25.

Eligibility:

CD25+ CTCL based on immunohistochemistry or flow cytometry of blood. Patients must have measurable stage 1b-IV disease which progressed after greater than or equal 2 prior systemic or topical therapies. Labs required: alanine aminotransferase (ALT) and aspartate aminotransferase (AST) less than or equal to 2.5-time upper limit, albumin greater than or equal 3, bilirubin less than or equal to 2.2, creatinine less than or equal to 2.0 (unless creatinine clearance greater than or equal to 50 ml/min), absolute neutrophil count (ANC) greater than or equal to 1000/ul, and platelets greater than or equal to 50,000/ul (ANC and platelets greater than or equal 500 and 10,000 if blood/marrow involvement).

Design:

Patients receive LMB-2 30 ug/Kg QOD time 3 every 4 weeks in absence of neutralizing antibodies or progressive disease. Dose escalation to 40 ug/Kg QOD times 3 if less than 2/6 dose limiting toxicity (DLT) at 30 ug/Kg times 3. 1st stage is 16 patients, to expand to 25 if greater than 1 of 16 patients respond.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients must have histopathological evidence of cluster of differentiation 25 (CD25) + cutaneous T-cell lymphoma (CTCL) confirmed by the National Institutes of Health (NIH) pathology department.

One of the following must be present:

Greater than or equal to 20 percent expression of CD25 on the lymphocytes in the skin at a site of a patch, plaque, or tumor.

Greater than or equal to 20 percent of the peripheral blood Sezary cells must be CD25+.

Measurable stage Ib-IV disease that has progressed after at least 2 prior systemic or topical therapies.

Patients must have a Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 2 and be at least 18 years old.

Patients must be able to understand and give informed consent.

Patients must be 4 weeks from any monoclonal antibodies.

Patients must be greater than or equal to 3 weeks from any CTCL-specific therapy and have evidence of progressive disease.

Patients who are on chronic steroids must be on a stable dose of Prednisone less than or equal to 20 mg/day (or equivalent dose of another steroid) for at least 3 weeks and have evidence of progressive disease.

Female patients of childbearing potential must have a negative pregnancy test and must use effective contraception (a barrier form of contraception).

The transaminases alanine aminotransferase (ALT) and aspartate aminotransferase (AST) must each be less than or equal to 2.5-times the upper limits of normal.

Albumin must be greater than or equal to 3.0 gm/dL.

Total bilirubin must be less than or equal to 2.2 mg/dL.

The creatinine must be less than or equal to 2.0 mg/dL or the creatinine clearance must be greater than or equal to 50 ml/min.

The absolute neutrophil count (ANC) must be greater than or equal to 1000/mm^3 and the unsupported platelet count must be greater than or equal to 50,000/mm^3 in patients without blood or bone marrow involvement.

If there is blood or bone marrow involvement, the ANC must be greater than or equal to 500 mm^3 and the platelets must be greater than or equal to 10,000/mm^3.

The cardiac ejection fraction as assessed by echocardiogram or nuclear medicine study must not be less than the institutional limit of normal.

Pulmonary function studies must demonstrate a carbon monoxide diffusing capacity (DLCO) greater than or equal to 55 percent and a forced expiratory volume 1 (FEV1) greater than or equal to 60 percent of normal for inclusion.

EXCLUSION CRITERIA:

Patients whose serum neutralizes LMB-2 in tissue culture, due either to anti-toxin or anti-mouse-IgG antibodies.

No patient whose serum neutralizes greater than 75 percent of the activity of 1 microg/mL of LMB-2 will be treated.

Patients who are pregnant or breast-feeding.

Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection,

symptomatic congestive heart failure,

unstable angina pectoris,

cardiac arrhythmia,

or psychiatric illness/social situations that would limit compliance with study requirements.

Patients who are human immunodeficiency virus (HIV) positive,

hepatitis B antigen positive,

hepatitis C polymerase chain reaction (PCR) positive,

or who have other chronic liver disease.

Patients with symptomatic cardiac or pulmonary disease.

Patients on warfarin therapy.

Such patients may be eligible if they can be switched to heparin or low-molecular weight heparin therapy and are off warfarin at least 4 days prior to study enrollment.

Active cancer requiring treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2004-04-30 (Actual); Primary Completion 2011-12-31 (Actual); Study Completion 2011-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Kreitman, M.D., Principal Investigator — National Cancer Institute, National Institutes of Health
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel RS, Pandolfino T, Guitart J, Rosen S, Kuzel TM. Primary cutaneous T-cell lymphoma: review and current concepts. J Clin Oncol. 2000 Aug;18(15):2908-25. doi: 10.1200/JCO.2000.18.15.2908. PMID 10920140
- [Background] Diamandidou E, Cohen PR, Kurzrock R. Mycosis fungoides and Sezary syndrome. Blood. 1996 Oct 1;88(7):2385-409. No abstract available. PMID 8839829
- [Background] Weinstock MA, Horm JW. Mycosis fungoides in the United States. Increasing incidence and descriptive epidemiology. JAMA. 1988 Jul 1;260(1):42-6. PMID 3379722
- [Derived] Matsushita K, Margulies I, Onda M, Nagata S, Stetler-Stevenson M, Kreitman RJ. Soluble CD22 as a tumor marker for hairy cell leukemia. Blood. 2008 Sep 15;112(6):2272-7. doi: 10.1182/blood-2008-01-131987. Epub 2008 Jul 2. PMID 18596230
- See also: International Workshop to Standardize Response Criteria for Non-Hodgkin's Lymphomas — http://ncbi.nlm.nih.gov/pubmed/10561185

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LMB-2 for Cutaneous Tcell Lymphoma
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | LMB-2 for Cutaneous Tcell Lymphoma
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.85 (17.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Response is assessed by the International Workshop's Response Criteria (IWRC) for Non-Hodgkin's Lymphomas which favors the sum of the bidimensional products for tumor measurements. Complete response is no evidence of disease. Complete response unconfirmed (CRu) is a complete response in every category except CRu in lymph nodes. Partial response is a partial response in every measurable category with non-progressive disease elsewhere. Progressive disease is progressive disease in every category. Stable disease is neither partial response nor progressive disease. For additional details about the IWRC see the protocol link module.
Time Frame: Patients were followed for at least 30 days after last treatment. Because the protocol allows 6 treatment cycles, this can be up to 7 months.
Measure: Number; unit: Participants
Arm/Group | LMB-2 for Cutaneous Tcell Lymphoma
Number analyzed (Participants) | 10
Participants
  Complete Response | 0
  Complete Response unconfirmed | 0
  Partial Response | 1
  Progressive Disease | 1
  Stable Disease | 8

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For the detailed list of adverse events see the adverse event module.
Time Frame: Date treatment consent signed to date off study, approximately 6 years, 8 months and 17 days.
Measure: Count of Participants; unit: Participants
Arm/Group | LMB-2 for Cutaneous Tcell Lymphoma
Number analyzed (Participants) | 10
Participants | 10

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 6 years, 8 months and 17 days.
Arm/Group | LMB-2 for Cutaneous Tcell Lymphoma
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 3/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LMB-2 for Cutaneous Tcell Lymphoma (N=10)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1 (1)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 1 (1)
Infection (documented clinically or microbiologically) (Infections and infestations) | 1 (1) — with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L):: Lung (pneumonia)
Infection with normal ANC or Grade 1 or 2 neutrophils::Bone (osteomyelitis) (Infections and infestations) | 1 (1)
CPK (creatine phosphokinase) (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LMB-2 for Cutaneous Tcell Lymphoma (N=10)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1 (1)
Hearing: patients with/without baseline auidgram and not enrolled in a monitoring program) (Ear and labyrinth disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
haptoglobin (Blood and lymphatic system disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 5 (9)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 2 (5)
Lymphopenia (Blood and lymphatic system disorders) | 4 (6)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1 (4)
Platelets (Blood and lymphatic system disorders) | 3 (4)
fibrinogen (Blood and lymphatic system disorders) | 1 (2)
PTT (Partial Thromboplastin Time) (Blood and lymphatic system disorders) | 2 (2)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 3 (3)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 7 (9)
Sweating (diaphoresis) (General disorders) | 1 (1)
Weight gain (General disorders) | 2 (2)
Weight loss (General disorders) | 1 (2)
Anorexia (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Distension/bloating, abdominal (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (2)
Hemorrhage, GU: Urinary NOS (Renal and urinary disorders) | 1 (1)
Hemorrhage/Bleeding - other (Specify) (General disorders) | 1 (1) — Hemorrhage of the feet
Infection with normal ANC or Grade 1 or 2 neutrophils::Catheter-related (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Conjunctiva (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Skin (cellulitis) (Infections and infestations) | 1 (1)
Edema: head and neck (Blood and lymphatic system disorders) | 1 (1)
Edema: limb (Blood and lymphatic system disorders) | 6 (8)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 4 (4)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 6 (9)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 6 (15)
Alkaline phosphatase (Metabolism and nutrition disorders) | 2 (2)
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 1 (2)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 1 (2)
CPK (creatine phosphokinase) (Metabolism and nutrition disorders) | 4 (10)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 1 (1)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 2 (4)
Creatinine (Metabolism and nutrition disorders) | 3 (5)
GGT (gamma-Glutamyl transpeptidase) (Metabolism and nutrition disorders) | 1 (1)
Hemoglobinuria (Metabolism and nutrition disorders) | 1 (1)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 1 (1)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 7 (9)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 1 (1)
Proteinuria (Metabolism and nutrition disorders) | 3 (3)
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 2 (2)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 3 (4)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 1 (1)
Confusion (Nervous system disorders) | 2 (2)
Neurology-Other (Specify, neurology: dizziness) (Nervous system disorders) | 1 (1)
Psychosis (hallucinations/delusions) (Nervous system disorders) | 1 (1)
Watery eye (epiphora, tearing) (Eye disorders) | 1 (1)
Pain::Chest wall (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pain::Head/headache (Nervous system disorders) | 2 (2)
Pain::Muscle (Musculoskeletal and connective tissue disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Pleural effusion/non-malignant (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Acute vascular leak syndrome (Vascular disorders) | 5 (5)
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2011-08-03): https://cdn.clinicaltrials.gov/large-docs/35/NCT00080535/Prot_SAP_ICF_001.pdf